CLINICAL TRIAL: NCT06766058
Title: Evaluating the Effectiveness of Aromatherapy for Alleviating Distress in Breast Cancer Patients Before Radiotherapy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ASTER 2
Record Dates: First submitted 2024-12-22; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Inhalation Aromatherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Carrier State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator)
  Interventions: Other: Carrier oil
- Intervention Group (Experimental)
  Interventions: Other: Asian plant extract blend

INTERVENTIONS:
Other: Carrier oil — Inhaler stick containing 2 drops of carrier oil.
  Arms: Control Group
Other: Asian plant extract blend — Inhaler stick containing 2 drops of Asian plant extract blend.
  Arms: Intervention Group

SUMMARY:
ASTER is a multi-part study that aims to prospectively establish evidence for the implementation of aromatherapy as complementary therapy within cancer care in the Singapore context. ASTER 2 study evaluates how extracts from Asian aromatic plants with familiar aromas introduced as inhalation therapy can alleviate distress in breast cancer patients scheduled to undergo radiotherapy (RT).

DETAILED DESCRIPTION:
On the day of CT Simulation, a research coordinator from the team will obtain consent from the eligible patients. Patient related outcomes will be collected from the consented patients. Study team will meet the patient 2 weeks later, on the day of their first radiotherapy session. Patient will be given an hour before the radiotherapy session begin. During this time distress score will be assessed, blood pressure and pulse rate will be measured, and saliva sample be collected. Patients will then be provided with the Inhaler stick containing 2 drops of either carrier oil (placebo), or Asian plant extract blend (intervention), which will be prepared prior to the study recruitment.

Patient will be instructed to hold the inhaler stick at about 8 cm (a hand fist's distance) away from their nose, to take up to 3 sniffs. This will be repeated with every 5 minutes of interval for 20 minutes of duration. After completion of the inhalation procedure, anxiety & distress score will be assessed, blood pressure and pulse rate will be measured, and saliva sample be collected.

A total of 300 breast cancer patients scheduled to undergo radiotherapy for the first time will be recruited in a randomized double-blind, 2-arm study: 150 patients in a Placebo-Control-Group, 150 patients in the Aromatherapy-Intervention-Group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 years old and above
2. Confirmed diagnosis of breast cancer of any stage
3. Scheduled to undergo radiotherapy for the first time
4. Capable of providing informed consent

Exclusion Criteria:

1. Physically or mentally incapable of providing verbal/written consent
2. Known or suspected hypersensitivity/allergy to essential oils or any components of the formulations
3. Airway hypersensitivity to fragrances, paint fumes or turpentine
4. Taking medications for anxiety (e.g. benzodiazepines) before radiotherapy
5. Pregnant, breastfeeding, or intending to conceive during study period

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The impact of Inhalation Aromatherapy Intervention on Distress. | Baseline (on CT Simulation Day), Before Intervention (on RT day), and After 20 minutes of Aromatherapy Intervention (on RT day).
  Changes of Distress Score (Distress Score from a scale of 0 - 10).
The impact of Inhalation Aromatherapy Intervention on Anxiety. | Baseline (on CT Simulation Day), After 20 minutes of Aromatherapy Intervention (on RT day).
  Change of General Anxiety Disorder Score (GAD-7 Score from a scale of 0 - 21) between Baseline and After Intervention.
The impact of Inhalation Aromatherapy Intervention on Cortisol (stress hormones). | Before Intervention (on RT day), After 20 minutes of Aromatherapy Intervention (on RT day).
  Change of Cortisol Levels in nmol/L between Before Intervention and After Intervention.

SECONDARY OUTCOMES:
The impact of Inhalation Aromatherapy Intervention on blood pressure. | Before Intervention (on RT day), After 20 minutes of Aromatherapy Intervention (on RT day).
  Change of blood pressure (in mmHg) between Before Intervention and After Intervention.
The impact of Inhalation Aromatherapy Intervention on pulse rate. | Before Intervention (on RT day), After 20 minutes of Aromatherapy Intervention (on RT day).
  Change of pulse rate (in bpm) between Before Intervention and After Intervention.
The safety outcomes associated with Inhalation Aromatherapy Intervention. | After 20 minutes of Aromatherapy Intervention (on RT day).
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Fuh-Yong Wong, MBBS, FRCR, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No